CLINICAL TRIAL: NCT06186349
Title: The Effect and Mechanism of Gene Variation on Neonatal Hyperbilirubinemia
Acronym: EMOGVONHB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, HaoHu, Project leader, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: EMGVNHB
Record Dates: First submitted 2023-12-13; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Neonatal Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Any newborn who joined the project, his/her parents will be informed and signed informed consent, in the newborn clinical treatment process to collect venous blood 2ml for gene sequencing and mutation screening
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- non-significant hyperbilirubinemia: including 500 cases of non-significant hyperbilirubinemia ( TSB / TCB < 205umol / L )
  Interventions: Genetic: Genomic sequencing
- significant hyperbilirubinemia: 500 cases of significant hyperbilirubinemia ( 205umol / L ≤ TSB / TCB < 342umol / L )
  Interventions: Genetic: Genomic sequencing
- severe hyperbilirubinemia: 500 cases of severe hyperbilirubinemia ( TSB / TCB ≥ 342umol / L )
  Interventions: Genetic: Genomic sequencing
- Extremely severe hyperbilirubinemia: 500 cases ( TSB / TCB ≥ 428umol / L )
  Interventions: Genetic: Genomic sequencing

INTERVENTIONS:
Genetic: Genomic sequencing — Newborns with neonatal hyperbilirubinemia who did not randomly receive genome sequencing will receive a Genomic Newborn Sequencing Report which will include pathogenic or likely pathogenic variants identified in genes associated with childhood-onset disease.

SUMMARY:
Neonatal hyperbilirubinemia ( NHB ) has many causes and is difficult to diagnose, and genetic factors play an important role in the metabolism of bilirubin. However, there is no literature report on the correlation between jaundice gene polymorphism and clinical manifestation polymorphism in big data population. This project intends to conduct a prospective observational study led by the Department of Pediatrics of the Sixth Affiliated Hospital of Sun Yat-sen University and in conjunction with a multi-center cooperative hospital : ( 1 ) A total of 2,000 NHB neonatal dry blood spot samples were included for 24 genetic screening tests for 29 NHB-related genetic diseases. The construction of the gene database was completed and the carrying and pathogenicity of NHB-related genes in the population was analyzed to provide a scientific basis for the selection of mutation sites for large-scale NHB gene screening ; ( 2 ) Collect neonatal clinical data and percutaneous bilirubin levels through the hospital inpatient system and the ' percutaneous jaundice meter home monitoring + software doctor-patient interconnection ' method, complete the construction of the intelligent NHB clinical database, and analyze the impact of jaundice-related genes on NHB ; ( 3 ) Integrated analysis to understand the differences in the carrying rate of pathogenic genes in different degrees and special types of jaundice, and to explore the differences in the degree of jaundice carrying single or multiple jaundice pathogenic genes. This study will evaluate the feasibility of jaundice gene screening program in the detection of jaundice-related inherited metabolic diseases, and provide a basis for early treatment and prevention of NHB.

DETAILED DESCRIPTION:
Adverse reactions: In this study, only 3 drops of neonatal heel peripheral blood were collected for genetic analysis and statistical analysis of percutaneous jaundice values. No human trials were involved. Family members were willing to know the genetic test results and the genetic test results were positive. Family members may have a certain psychological burden. We will provide free professional genetic counseling, as detailed as possible to inform the hazards of this genetic defect, treatment and other related information to help. Psychiatrists can be arranged for free psychological counseling if necessary.

Ethical approval: This clinical study follows the Helsinki Declaration ( 2013 edition ), the ethical principles of human medical research and the relevant clinical research norms and regulations in China.

This clinical study was approved by the Research Ethics Committee / Institutional Review Boards ( REC/IRBs ).

This clinical study is an observational clinical study initiated by researchers. The clinical research protocol ( including informed consent and case report forms, etc. ) and other information provided to the family members or guardians of the newborn were reviewed and approved by the ethics committee of the clinical research team leader unit and the participating units.

Informed consent: Before the start of the clinical study, the researchers completely and comprehensively introduced the purpose, process, method, and the interests and risks of the newborn to the parents or legal representatives who met the inclusion criteria. A written informed consent form was given to each parent or guardian of the newborn before enrollment, so that he / she had sufficient time to consider whether to consent to the collection of neonatal information to participate in this clinical study. After obtaining the informed consent of each newborn 's parent or legal representative and signing the informed consent form, researchers can begin to collect relevant data.

Privacy protection: All members of the research team, including the primary researchers and their authorized researchers, must comply with all local and regional regulatory requirements and applicable privacy regulations.

Each newborn participating in this study will be assigned a unique number and an institutional identifier.

All research data will be stored in a confidential electronic system and stored for at least 3 years after the completion of the study.

The coding table for recording neonatal information and research will be kept by the researcher (PI) in a locked file cabinet or in a password-protected database. Only researchers and their authorized researchers have the right to access the coding table.

The coding table that records the name of the hospital and the institution identification number will be saved by the research team in a locked file cabinet, which is only limited to access by limited research members. The identity of each subject of observation should be kept confidential in research reports and related publications.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-28 days
* gestational age ≥ 35 weeks
* Birth weight ≥ 2.5 kg and < 4 kg.

Exclusion Criteria:

* Neonatal data with unclear clinical basic information ;
* Lack of traceability core information data ;
* data that the test results cannot be analyzed and interpreted ;
* Sample collection is not qualified and unwilling to cooperate with re-sampling.
* Newborns with severe deformity and severe lethal inherited metabolic diseases

Ages: 1 Day to 28 Days | Sex: All
Age Groups: Child
Study Population: This study is a prospective observational study. According to the positive mutation rate of NHB-related genes in neonatal hyperbilirubinemia, P is about 30 %, the test level α = 0.05 and the allowable error δ = 2 %, n ( sample size ) = ( Uα / δ ) 2 * p * ( 1-P ) ≈ 2000 cases. A total of 2000 neonates were included, including 500 cases of non-significant hyperbilirubinemia ( TSB / TCB < 205umol / L ) ; ( 2 ) 500 cases of significant hyperbilirubinemia ( 205umol / L ≤ TSB / TCB < 342umol / L ) ; ( 3 ) 500 cases of severe hyperbilirubinemia ( TSB / TCB ≥ 342umol / L ) ; (4) Extremely severe hyperbilirubinemia 500 cases ( TSB / TCB ≥ 428umol / L ).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of gene sequencing data in neonatal gene bank | From birth to completion of genetic screening, the process last up to 3 months.
  Each newborn that was sequenced was counted as 1. Keep all the data in the gene bank, and finally calculate the number of completed gene sequencing data.
Gene mutation rate | From birth to completion of genetic screening, the process last up to 3 months.
  Taking the number of newborn babies as denominator and the number of neonates with gene mutation detected in gene sequencing as molecules, the whole neonatal gene mutation rate in China was obtained.
carrying rate of pathogenic genes | From birth to completion of genetic screening, the process last up to 3 months.
  the carrying rate of pathogenic genes of common hereditary jaundice diseases in newborns was counted
phenotypic polymorphism | From birth to completion of genetic screening, the process last up to 3 months.
  analyze the correlation between gene polymorphism and clinical manifestations ( phenotypic polymorphism ) of neonatal hyperbilirubinemia.

CONTACTS AND LOCATIONS:
Overall Officials: Hu Hao, Study Director — Department of Pediatrics, The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, China
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu J, Lu AD, Zhang LP, Zuo YX, Jia YP. [Study of clinical outcome and prognosis in pediatric core binding factor-acute myeloid leukemia]. Zhonghua Xue Ye Xue Za Zhi. 2019 Jan 14;40(1):52-57. doi: 10.3760/cma.j.issn.0253-2727.2019.01.010. Chinese. PMID 30704229
- [Result] Olusanya BO, Kaplan M, Hansen TWR. Neonatal hyperbilirubinaemia: a global perspective. Lancet Child Adolesc Health. 2018 Aug;2(8):610-620. doi: 10.1016/S2352-4642(18)30139-1. Epub 2018 Jun 28. PMID 30119720
- [Result] Watchko JF, Lin Z. Exploring the genetic architecture of neonatal hyperbilirubinemia. Semin Fetal Neonatal Med. 2010 Jun;15(3):169-75. doi: 10.1016/j.siny.2009.11.003. Epub 2009 Dec 21. PMID 20022574
- [Result] Yang H, Wang Q, Zheng L, Zheng XB, Lin M, Zhan XF, Yang LY. Clinical Significance of UGT1A1 Genetic Analysis in Chinese Neonates with Severe Hyperbilirubinemia. Pediatr Neonatol. 2016 Aug;57(4):310-7. doi: 10.1016/j.pedneo.2015.08.008. Epub 2015 Dec 2. PMID 26727668

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT06186349/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT06186349/ICF_001.pdf